CLINICAL TRIAL: NCT03371823
Title: Losartan and ET-1 Mediated Constriction in Postmenopausal Women With High Blood Pressure
Brief Title: Vascular Dysfunction in Hypertensive Postmenopausal Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We experienced challenges recruiting unmedicated women with high blood pressure for the intervention.
Sponsor: University of Delaware (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Megan M. Wenner, Assistant professor, University of Delaware
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1009297
Record Dates: First submitted 2017-11-22; First posted 2017-12-13 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: Hypertension; Endothelin-1 receptor
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normotensive (Other): Normotensive PMW will complete an experimental visit to assess vascular function. All women will wear an ambulatory BP monitor during the 24 hours preceding the experimental visit to confirm BP classification. Large blood vessel function will be assessed using two non-invasive techniques: 1. Flow Mediated Dilation (FMD) 2. Pulse Wave Analysis and Pulse Wave Velocity. ET-1 mediated vasoconstrictor tone is assessed by measuring the cutaneous blood flow during microdialysis perfusions of ET-A and ET-B receptor antagonist. ET-1 production, ET-A and ET-B receptor expression is assessed from antecubital vein endothelial cells and skin punch biopsy samples.
  Interventions: Other: Normotensive
- Hypertensives (Experimental): Hypertensive women will be tested at baseline and then administered Losartan 50 mg once a day at night for 14 days. Vascular function is measured at baseline and again after 2 weeks of losartan. All women will wear an ambulatory BP monitor during the 24 hours preceding the experimental visits to confirm BP classification. Large blood vessel function will be assessed using two non-invasive techniques: 1. Flow Mediated Dilation (FMD) 2. Pulse Wave Analysis and Pulse Wave Velocity. ET-1 mediated vasoconstrictor tone is assessed by measuring the cutaneous blood flow during microdialysis perfusions of ET-A and ET-B receptor antagonist. ET-1 production, ET-A and ET-B receptor expression is assessed from antecubital vein endothelial cells and skin punch biopsy samples.
  Interventions: Drug: Hypertensives

INTERVENTIONS:
Other: Normotensive — FMD is a measure of endothelial function by assessing the degree to which vessel dilates in response to increased flow. Pulse Wave Analysis and Pulse Wave Velocity assesses arterial stiffness and wave reflection in all women. Laser Doppler flowmetry is used in combination with cutaneous microdialysis as a minimally invasive technique to examine mechanisms of vascular function. ET-B and ET-A receptor antagonists will be perfused via intradermal microdialysis fibers while measuring cutaneous blood flow. ET-1 production and ET-B receptor expression in endothelial cells collected from an antecubital vein will also be assessed. Immunohistochemistry will be performed on skin punch biopsy samples to assess for protein expression of ET-A and ET-B receptors.
  Arms: Normotensive
Drug: Hypertensives — ANG II increases the synthesis of ET-1 and alters ET-A/B receptor expression, thus affecting ET-1 bioavailability. Losartan is an ANG II receptor antagonist which attenuates ET-1 production. Losartan 50 mg daily is administered for 14 days to hypertensive women. FMD is used to measure endothelial function. Pulse Wave Analysis and Pulse Wave Velocity assesses arterial stiffness and wave reflection. Laser Doppler flowmetry with cutaneous microdialysis is used to examine vascular function when ET-A and ET-B receptor antagonists is perfused via intradermal microdialysis fibers. ET-1 production and ET-B receptor expression in endothelial cells collected from an antecubital vein will be assessed. Skin punch biopsy samples will be used to assess for protein expression of ET-A and ET-B receptors.
  Arms: Hypertensives

SUMMARY:
The purpose of this study is to investigate the role of ET-1 in mediating vasoconstrictor tone in hypertensive postmenopausal women (PMW) alone and in combination with a commonly prescribed Angiotensin II (ANG II) antagonist. The long term goal is to understand the mechanisms contributing to hypertension (HTN) in PMW. This study is the first step in reaching our goal.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in women, and mortality from CVD is higher in PMW compared to age-matched men. PMW are at a greater risk for developing HTN, a major risk factor for CVD. They are also more likely to have uncontrolled or resistant HTN despite medication.

ANG II is a common therapeutic target for the treatment HTN. ANG II blockade is highly effective in normalizing blood pressure (BP) in hypertensive male rats, but does not reduce BP to the same degree in hypertensive post menopausal female rats. Endothelin-1 (ET-1) receptor antagonists reduce BP in hypertensive postmenopausal female rats, but have no effect on males. Thus the mechanisms contributing to HTN in female rats and likely women, particularly after menopause, are complex, multifactorial and not completely understood.

After menopause, the vasoconstrictor effects of both ANG II and ET-1 are amplified in animal models. As such, these two predominant pathways may contribute to the high incidence of HTN in PMW. ET-1 is a potent vasoconstrictor produced and released by endothelial cells that binds to two receptor subtypes, ET-A and ET-B. While both receptors are located on vascular smooth muscle (VSM) and mediate vasoconstriction, ET-B receptors are also located on the endothelium and mediate vasodilation via nitric oxide.

Importantly, the production of ET-1 and expression of ET-A and B receptors can be modulated by hormones such as estradiol and ANG II. Estradiol attenuates ET-1 production, and reduces ET-1 mediated vasoconstriction via an ET-B receptor mechanism in vitro. Thus, decline in estradiol after menopause may enhance vasoconstrictor tone via ET-1 and lead to HTN. ET-1 also potentiates the vasoconstrictor effects of ANG II since the vasoconstrictor and hypertensive effects of ANG II are ameliorated by ET-1 receptor blockade. Additionally, ANG II stimulates the synthesis of ET-1 and upregulates ET-A and ET-B receptor expression on VSM. The ANG II receptor antagonist Losartan reduces ET-A and ET-B receptor expression and attenuates the constrictor effects of ET-1 in a diabetic rat model. Therefore, ET-1 is an important independent factor contributing to HTN in PMW, but therapeutic agents targeting both ANG II and ET-1 may have greater efficacy given their interactions.

The investigators propose a comprehensive assessment of vascular function by measuring blood flow responses in the cutaneous circulation during perfusion of ET-1 receptor antagonists via microdialysis, combined with measures of intracellular protein and receptor expression of endothelial cells and skin punch biopsies collected from normotensive and hypertensive PMW. Investigators central hypothesis is that hypertensive PMW have greater ET-1 mediated vasoconstrictor tone due to increased ET-1 expression, down-regulation of ET-B receptors on endothelial cells and up-regulation of both ET-A and ET-B receptors on VSM leading to increased vasoconstriction and HTN. Investigators further hypothesize that ANG II exacerbates the increase in ET-1, and ET-A and ET-B receptor expression contributing to exaggerated constriction with HTN in PMW.

ELIGIBILITY:
Inclusion Criteria: - Women.

* > 1year post menopausal.
* Age range 50-70 years
* Resting ECG in normal limits
* Standard blood chemistry within normal limits
* Systolic blood pressure: <130mm Hg for normotensives; >130mm Hg for hypertensives.
* Diastolic blood pressure: < 80mm Hg for normotensives; > 80mm Hg for hypertensives.

Exclusion Criteria:

* History of cardiovascular disease
* Blood clots or stroke
* Cancer
* Diabetes
* Kidney or Liver disease
* Obesity (BMI>35kg/m2)
* Pregnant/Breast feeding
* Current use of hormone therapy
* Current use of tobacco products
* High cholesterol
* Current use of anti-hypertensive meds

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Wenner, Ph.D, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Background] Barton M, Meyer MR. Postmenopausal hypertension: mechanisms and therapy. Hypertension. 2009 Jul;54(1):11-8. doi: 10.1161/HYPERTENSIONAHA.108.120022. Epub 2009 May 26. No abstract available. PMID 19470884
- [Background] Kim JK, Alley D, Seeman T, Karlamangla A, Crimmins E. Recent changes in cardiovascular risk factors among women and men. J Womens Health (Larchmt). 2006 Jul-Aug;15(6):734-46. doi: 10.1089/jwh.2006.15.734. PMID 16910905
- [Background] Yanes LL, Romero DG, Iles JW, Iliescu R, Gomez-Sanchez C, Reckelhoff JF. Sexual dimorphism in the renin-angiotensin system in aging spontaneously hypertensive rats. Am J Physiol Regul Integr Comp Physiol. 2006 Aug;291(2):R383-90. doi: 10.1152/ajpregu.00510.2005. Epub 2006 Mar 30. PMID 16914423
- [Background] Yanes LL, Romero DG, Iliescu R, Zhang H, Davis D, Reckelhoff JF. Postmenopausal hypertension: role of the Renin-Angiotensin system. Hypertension. 2010 Sep;56(3):359-63. doi: 10.1161/HYPERTENSIONAHA.110.152975. Epub 2010 Aug 2. PMID 20679182
- [Background] Reckelhoff JF. Gender differences in the regulation of blood pressure. Hypertension. 2001 May;37(5):1199-208. doi: 10.1161/01.hyp.37.5.1199. PMID 11358929
- [Background] Yanes LL, Reckelhoff JF. Postmenopausal hypertension. Am J Hypertens. 2011 Jul;24(7):740-9. doi: 10.1038/ajh.2011.71. Epub 2011 Apr 21. PMID 21509049
- [Background] Yanes LL, Romero DG, Cucchiarelli VE, Fortepiani LA, Gomez-Sanchez CE, Santacruz F, Reckelhoff JF. Role of endothelin in mediating postmenopausal hypertension in a rat model. Am J Physiol Regul Integr Comp Physiol. 2005 Jan;288(1):R229-33. doi: 10.1152/ajpregu.00697.2003. Epub 2004 Aug 19. PMID 15319224
- [Background] Lima R, Yanes LL, Davis DD, Reckelhoff JF. Roles played by 20-HETE, angiotensin II and endothelin in mediating the hypertension in aging female spontaneously hypertensive rats. Am J Physiol Regul Integr Comp Physiol. 2013 Feb;304(3):R248-51. doi: 10.1152/ajpregu.00380.2012. Epub 2012 Dec 5. PMID 23220478
- [Background] Haynes WG. Endothelins as regulators of vascular tone in man. Clin Sci (Lond). 1995 May;88(5):509-17. doi: 10.1042/cs0880509. PMID 7614809
- [Background] Ishikawa K, Ihara M, Noguchi K, Mase T, Mino N, Saeki T, Fukuroda T, Fukami T, Ozaki S, Nagase T, et al. Biochemical and pharmacological profile of a potent and selective endothelin B-receptor antagonist, BQ-788. Proc Natl Acad Sci U S A. 1994 May 24;91(11):4892-6. doi: 10.1073/pnas.91.11.4892. PMID 8197152
- [Background] Yanagisawa M, Kurihara H, Kimura S, Tomobe Y, Kobayashi M, Mitsui Y, Yazaki Y, Goto K, Masaki T. A novel potent vasoconstrictor peptide produced by vascular endothelial cells. Nature. 1988 Mar 31;332(6163):411-5. doi: 10.1038/332411a0. PMID 2451132
- [Background] Juan SH, Chen JJ, Chen CH, Lin H, Cheng CF, Liu JC, Hsieh MH, Chen YL, Chao HH, Chen TH, Chan P, Cheng TH. 17beta-estradiol inhibits cyclic strain-induced endothelin-1 gene expression within vascular endothelial cells. Am J Physiol Heart Circ Physiol. 2004 Sep;287(3):H1254-61. doi: 10.1152/ajpheart.00723.2003. Epub 2004 May 6. PMID 15130882
- [Background] Pedersen SH, Nielsen LB, Mortensen A, Nilas L, Ottesen B. Progestins oppose the effects of estradiol on the endothelin-1 receptor type B in coronary arteries from ovariectomized hyperlipidemic rabbits. Menopause. 2008 May-Jun;15(3):503-10. doi: 10.1097/gme.0b013e318156f803. PMID 18188139
- [Background] Wenzel RR, Ruthemann J, Bruck H, Schafers RF, Michel MC, Philipp T. Endothelin-A receptor antagonist inhibits angiotensin II and noradrenaline in man. Br J Clin Pharmacol. 2001 Aug;52(2):151-7. doi: 10.1046/j.0306-5251.2001.01422.x. PMID 11488771
- [Background] Gossl M, Mitchell A, Lerman A, Opazo Saez A, Schafers RF, Erbel R, Philipp T, Wenzel RR. Endothelin-B-receptor-selective antagonist inhibits endothelin-1 induced potentiation on the vasoconstriction to noradrenaline and angiotensin II. J Hypertens. 2004 Oct;22(10):1909-16. doi: 10.1097/00004872-200410000-00013. PMID 15361762
- [Background] Ballew JR, Fink GD. Role of ET(A) receptors in experimental ANG II-induced hypertension in rats. Am J Physiol Regul Integr Comp Physiol. 2001 Jul;281(1):R150-4. doi: 10.1152/ajpregu.2001.281.1.R150. PMID 11404288
- [Background] Barton M, Shaw S, d'Uscio LV, Moreau P, Luscher TF. Angiotensin II increases vascular and renal endothelin-1 and functional endothelin converting enzyme activity in vivo: role of ETA receptors for endothelin regulation. Biochem Biophys Res Commun. 1997 Sep 29;238(3):861-5. doi: 10.1006/bbrc.1997.7394. PMID 9325182
- [Background] Dimitrijevic I, Edvinsson ML, Chen Q, Malmsjo M, Kimblad PO, Edvinsson L. Increased expression of vascular endothelin type B and angiotensin type 1 receptors in patients with ischemic heart disease. BMC Cardiovasc Disord. 2009 Aug 25;9:40. doi: 10.1186/1471-2261-9-40. PMID 19706169
- [Background] Kanno K, Hirata Y, Tsujino M, Imai T, Shichiri M, Ito H, Marumo F. Up-regulation of ETB receptor subtype mRNA by angiotensin II in rat cardiomyocytes. Biochem Biophys Res Commun. 1993 Aug 16;194(3):1282-7. doi: 10.1006/bbrc.1993.1962. PMID 8352786
- [Background] Moreau P, d'Uscio LV, Shaw S, Takase H, Barton M, Luscher TF. Angiotensin II increases tissue endothelin and induces vascular hypertrophy: reversal by ET(A)-receptor antagonist. Circulation. 1997 Sep 2;96(5):1593-7. doi: 10.1161/01.cir.96.5.1593. PMID 9315552
- [Background] Kobayashi T, Nogami T, Taguchi K, Matsumoto T, Kamata K. Diabetic state, high plasma insulin and angiotensin II combine to augment endothelin-1-induced vasoconstriction via ETA receptors and ERK. Br J Pharmacol. 2008 Dec;155(7):974-83. doi: 10.1038/bjp.2008.327. Epub 2008 Aug 18. PMID 19029977
- [Background] Hong HJ, Chan P, Liu JC, Juan SH, Huang MT, Lin JG, Cheng TH. Angiotensin II induces endothelin-1 gene expression via extracellular signal-regulated kinase pathway in rat aortic smooth muscle cells. Cardiovasc Res. 2004 Jan 1;61(1):159-68. doi: 10.1016/j.cardiores.2003.10.019. PMID 14732213
- [Background] Kohno M, Horio T, Ikeda M, Yokokawa K, Fukui T, Yasunari K, Kurihara N, Takeda T. Angiotensin II stimulates endothelin-1 secretion in cultured rat mesangial cells. Kidney Int. 1992 Oct;42(4):860-6. doi: 10.1038/ki.1992.361. PMID 1333547
- [Background] Wenner MM, Sebzda KN, Kuczmarski AV, Pohlig RT, Edwards DG. ETB receptor contribution to vascular dysfunction in postmenopausal women. Am J Physiol Regul Integr Comp Physiol. 2017 Jul 1;313(1):R51-R57. doi: 10.1152/ajpregu.00410.2016. Epub 2017 Apr 24. PMID 28438762

RESULTS

PARTICIPANT FLOW:
Groups:
- Normotensive: Normotensive postmenopausal women (PMW) will complete an experimental visit to assess vascular function. All women will wear an ambulatory BP monitor during the 24 hours preceding the experimental visit to confirm BP classification. Large blood vessel function will be assessed using two non-invasive techniques: 1. Flow Mediated Dilation (FMD) 2. Pulse Wave Analysis and Pulse Wave Velocity. Endothelin-1 (ET-1) mediated vasoconstrictor tone is assessed by measuring the cutaneous blood flow during microdialysis perfusions of ET-A and ET-B receptor antagonist. ET-1 production, ET-A and ET-B receptor expression is assessed from antecubital vein endothelial cells and skin punch biopsy samples.
  Normotensive: FMD is a measure of endothelial function by assessing the degree to which vessel dilates in response to increased flow. Pulse Wave Analysis and Pulse Wave Velocity assesses arterial stiffness and wave reflection in all women. Laser Doppler flowmetry is used in combination with cutaneous microdialysis as a minimally invasive technique to examine mechanisms of vascular function. ET-B and ET-A receptor antagonists will be perfused via intradermal microdialysis fibers while measuring cutaneous blood flow. ET-1 production and ET-B receptor expression in endothelial cells collected from an antecubital vein will also be assessed. Immunohistochemistry will be performed on skin punch biopsy samples to assess for protein expression of ET-A and ET-B receptors.
Period: Overall Study
Arm/Group | Normotensive | Hypertensives
Started | 8 | 0 (We had trouble enrolling naive to therapy women with high blood pressure)
Completed | 7 | 0
Not Completed | 1 | 0
Not completed — Screen fail (did not meet inclusion criteria) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Normotensive BP <130/80mmHg Hypertensive BP >130/80mmHg
Groups:
- Total: Total of all reporting groups
Arm/Group | Normotensive | Hypertensives | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 0 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: ET-1 Mediated Constriction
Description: Cutaneous blood flow is measured via laser Doppler flowmetry during cutaneous microdialysis perfusions of ET-A and ET-B receptor antagonists as previously described by Wenner MM in 2017(see reference list).
Time Frame: Each participant was assessed at baseline and 2 weeks later.
Population: We were not able to recruit any hypertensive women naive to therapy for this arm of the study
Measure: Mean (Standard Error); unit: % change blood flow flux
Arm/Group | Normotensive | Hypertensives
Number analyzed (Participants) | 6 | 0
% change blood flow flux
  ETA blockade | 437 (999) |
  ETB blockade | 42 (14) |

2. Secondary Outcome: Endothelin Receptor A and B Expression
Description: ET-A and ET-B receptors will be examined using immunocytochemistry from 3mm skin punch biopsy in women pre/post losartan administration. This Secondary aim was not complete due to difficulty with enrollment (no data collected in these groups).
Time Frame: Baseline and 2 weeks later
Population: Due to difficulty with enrollment we were not able to complete this outcome
Arm/Group | Normotensive | Hypertensives
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline and 2 weeks later
Description: Standard definitions were used. No Adverse Events occurred.
Arm/Group | Normotensive | Hypertensives
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/0

LIMITATIONS AND CAVEATS:
We were not able to enroll naive to therapy hypertensive women for the Losartan arm of the trial and do not have data on this arm of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03371823/Prot_SAP_003.pdf
  • Informed Consent Form (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03371823/ICF_002.pdf